CLINICAL TRIAL: NCT06319209
Title: Timing of Surgery and the Evolution of Postoperative Outcomes in Breast Cancer Patients Undergoing Surgical Intervention Following Recovery From SARS-CoV-2 Infection: a Matched, Longitudinal, Prospective Cohort Study
Brief Title: Timing of Surgery and the Evolution of Postoperative Outcomes in Breast Cancer Patients Undergoing Surgical Intervention Following Recovery From SARS-CoV-2 Infection
Status: Active, not recruiting | Type: Observational
Sponsor: Fujian Medical University Union Hospital (Other)
Responsible Party: Principal Investigator, Chuan Wang, Head of Department of Breast Surgery, Fujian Medical University Union Hospital
Other Study IDs: 2024KY023
Record Dates: First submitted 2024-03-13; First posted 2024-03-19 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer; COVID-19; Postoperative Complications
MeSH Terms: conditions — Breast Neoplasms; COVID-19; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preoperative resolved COVID-19: Patients who had a history of SARS-CoV-2 infection prior to surgery underwent limited breast cancer operations in the Breast Surgery Department of our hospital after recovering from SARS-CoV-2 infection between January 2023 and March 2023.
  Interventions: Other: Preoperative resolved COVID-19
- Preoperative COVID-19 negative: Patients undergoing limited surgery for breast cancer in our Breast Surgery Department between June and August 2022 had no history of SARS-CoV-2 infection prior to surgery. However, they were diagnosed with COVID-19 after the first tumor evaluation following surgery, which occurred at least 90 days after the surgery.

INTERVENTIONS:
Other: Preoperative resolved COVID-19 — We observed postoperative outcomes only in patients who had or did not have COVID-19 before surgery, without any additional intervention.
  Groups: Preoperative resolved COVID-19

SUMMARY:
Perioperative SARS-CoV-2 infection significantly increases the risk of postoperative complications and mortality, while also exerting long-lasting impacts on multiple organs and systems. Due to the curtailment or cessation of non-emergency surgeries during the initial phase of the pandemic, there is a lack of evidence regarding the optimal timing and medium- to long-term postoperative outcomes of surgical intervention in breast cancer patients with prior SARS-CoV-2 infection, particularly after vaccination. We aim to investigate whether prior SARS-CoV-2 infection increases the risk of postoperative adverse outcomes in breast cancer patients and determine the optimal timing for surgical intervention during the pandemic, as well as to longitudinally assess the evolution of postoperative adverse outcomes within one year after COVID-19 and identify associated risk factors.

DETAILED DESCRIPTION:
This study employs a prospective cohort design with longitudinal and matched characteristics, focusing on breast cancer patients who underwent surgery after recovering from SARS-CoV-2 infection. Patients were stratified by the time of surgery relative to COVID-19 diagnosis. The Inverse Probability of Treatment Weighting (IPTW) method was used to match a control group (COVID-19 negative) based on patient, tumor, and surgical factors in order to compare composite indicators (including death, pneumonia, thrombosis, cardiac complications, and unplanned hospitalization) for evaluating the optimal timing of surgery. We investigated the longitudinal evolution of postoperative adverse outcomes and identified the relevant risk factors through logistic regression analysis.

ELIGIBILITY:
Inclusion Criteria:

* Breast cancer patients who underwent surgery after recovering from SARS-CoV-2 infection
* Breast cancer patients who had never been infected with SARS-CoV-2 before surgery

Exclusion Criteria:

* Distant metastasis
* Pregnancy-associated breast cancer
* Incomplete follow-up information

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The first group was the resolved COVID-19 group, which served as the experimental group and included patients who had recovered from SARS-CoV-2 infection between January 2023 and March 2023 and underwent limited breast cancer operations in our Breast Surgery Department. These patients had a history of SARS-CoV-2 infection before surgery. The second group was the pre-COVID-19 group, which served as the control group and included patients who underwent limited breast cancer operations in our Breast Surgery Department between June and August 2022 and had no history of SARS-CoV-2 infection before surgery. However, these patients were diagnosed with COVID-19 after the first tumor assessment after surgery (at least 90 days after surgery) and excluded patients who had been infected with SARS-CoV-2 within 90 days after surgery or showed distant metastases.
Sampling Method: Non-Probability Sample
Enrollment: 392 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
30-day postoperative outcomes | Within 30 days after surgery
  Composite indicators (including death, pneumonia, thrombosis, cardiac complications, and unplanned hospitalization) of COVID-19-related adverse outcomes within 30 days after surgery

SECONDARY OUTCOMES:
Postoperative outcomes at the time of the initial tumor assessment after surgery | The time of the initial tumor assessment after surgery (about 90 days after surgery)
  Composite indicators (including death, pneumonia, thrombosis, cardiac complications, and unplanned hospitalization) of COVID-19-related adverse outcomes at the time of the initial tumor assessment after surgery
12-month postoperative outcomes | Within 12 months after surgery
  Composite indicators (including death, pneumonia, thrombosis, cardiac complications, and unplanned hospitalization) of COVID-19-related adverse outcomes at 12 months after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Chuan Wang, Study Chair — Fujian Medical University Union Hospital
Locations (1):
- Fujian Medical University Union Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No